CLINICAL TRIAL: NCT06935253
Title: Towards Bridging Generalists to Subspecialists With Large Language Models
Brief Title: Large Language Models To Improve the Quality of Care of Cardiology Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Google LLC. (Industry)
Responsible Party: Principal Investigator, Jack O'Sullivan, Postdoctoral Fellow, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 78695
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hypertrophic Cardiomyopathy (HCM); Cardiomyopathy; Genetic Disease; Cardiology
Keywords: Large language models; Cardiology
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathies; Genetic Diseases, Inborn | interventions — Large Language Models

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluation of responses will be performed by assessors blinded to participant identity and treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Large Language Model (Active Comparator): This group will be given access to a Large Language Model
  Interventions: Other: Large Language Model
- Usual resources (No Intervention): Group will not be given access to a Large Language Model but will be encouraged to use any resources they usually use in their practice besides large language models (UpToDate, Dynamed etc).

INTERVENTIONS:
Other: Large Language Model — The intervention is a Large Language Model.
  Other Names: AMIE (Articulate Medical Intelligence Explorer)
  Arms: Large Language Model

SUMMARY:
This study evaluates the impact of large language models (LLMs) versus traditional decision support tools on clinical decision-making in cardiology. General cardiologists will be randomized to manage real patient cases from a cardiovascular genetic cardiomyopathy clinic, with or without AI assistance. Each case will be assessed by two cardiologists, and their responses will be graded by blinded subspecialty experts using a standardized evaluation rubric.

DETAILED DESCRIPTION:
Large language models have been shown to improve physician performance in simulated settings. Large language models have demonstrated promise in various healthcare contexts, including medical note-writing, addressing patient inquiries, and facilitating medical consultation. However, it remains uncertain whether large language models improve clinical reasoning of clinicians using real world cases.

Clinicians dedicate years of training to develop expertise, with clinical knowledge a key component. Clinicians have different areas of expertise, from generalists spanning diseases of all organ systems and patients of all ages, to subspecialists dedicated to often a handful of diseases effecting a specific organ. Both skill sets are vital to a well-functioning medical system, as generalists generally care for patients and refer to specialists when dedicated, specialty knowledge is required. There is a paucity of specialists, and thus the quality of triaging and referral to specialists is of upmost importance. We hypothesis that large language models may be able help generalists management complex patients, and improve their triage to specialists and subspecialists.

The scarcity of subspecialist medical expertise, particularly in rare, complex and life-threatening diseases, poses a significant challenge for healthcare delivery. This issue is particularly acute in cardiology where timely, accurate management determines outcomes. In this study, we will recruit General Cardiologists as participants who will be randomized to answer clinical management cases with or without access to a large language model. Each case is a real patient case of a patient referred to a subspeciality cardiovascular genetic cardiomyopathy clinic. Each case will be performed by two general cardiologists (one with access to a large language model and one without access). Each case has multiple components, and the participants will be asked to answer questions related to the management. Answers will be graded by independent, blinded subspeciality Cardiologists with expertise and training in genetic cardiomyopathies. An evaluation rubric was developed by 10 expert discussants.

ELIGIBILITY:
Inclusion Criteria:

* Board certified or board eligible Cardiologist.

Exclusion Criteria:

* Not currently practicing clinically

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Subspecialist Preference | Subspecialist evaluation will occur within 1 month of participant completing their assessment
  The primary outcome is the preference of the subspecialist between answers provided by a) Cardiologist with access to Large Language Model vs. b) Cardiologist without access to Large Language Model.

SECONDARY OUTCOMES:
Participants perspective on use of Large Language model | Within one-hour
  Percentage of Cardiologists that felt the use of the Large Language Model helped their assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Euan A Ashley, BSc, MB ChB, DPhil, Principal Investigator — Stanford University
Locations (1):
- Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The patient cases that will be used in this study will be deidentified and made publicly available. The code to conduct the statistical analysis will also be made available.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The deidentified patient cases and statistical analysis code will be made available within 6 months of study completion.
Access Criteria: It will be made publicly available and accessible by all.
URL: https://redivis.com/datasets/1z3x-2354972da?v=next